CLINICAL TRIAL: NCT06949605
Title: Quantitative Xylazine Measurement Among Non-Fatal Opioid Overdose Patients in the Emergency Department
Brief Title: Quantitative Xylazine Measurement in ED
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Love, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-24-01068; 5R25DA058490-02 (NIH)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Opioid Overdose; Substance Use Disorders
Keywords: Opioid; Xylazine; Substance Use
MeSH Terms: conditions — Opiate Overdose; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine and Waste Blood/Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Opioid Overdose: Individuals presenting to the ED with a suspected Opioid Overdose with Xylazine exposure.

SUMMARY:
Quantitative Xylazine Measurement Among Non-Fatal Opioid Overdose (OD) Patients in the Emergency Department (ED)

DETAILED DESCRIPTION:
Xylazine, a veterinary medication and alpha-2 agonist drug with clinical effects including prolonged sedation and skin/soft tissue wounds, has been increasingly detected with fentanyl in the illicit opioid supply. Due to its rapid emergence, limited knowledge exists regarding xylazine's health effects. In this proposed research, Dr. Love will measure xylazine and its metabolites in blood and urine samples using laboratory and point-of-care assays. Working at two New York City emergency departments, Dr. Love will collect waste serum and urine from opioid overdose patients to measure xylazine and its metabolite concentrations. The researcher will also perform qualitative assessment of urine samples with xylazine test strips to characterize urine xylazine detection using a harm reduction tool.

ELIGIBILITY:
Inclusion Criteria:

* ED patient
* Opioid OD (both NPS and non-NPS)
* Availability of waste blood specimens for analysis
* Availability of waste urine specimens for analysis

Exclusion Criteria:

- Children under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participating sites will enroll all opioid ODs presenting to Mount Sinai Hospital and Elmhurst Hospital Emergency Departments, regardless of whether or not a consultation by a medical toxicologist was requested (i.e., all consecutive opioid ODs).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Xylazine Concentration in Blood | 6 months
  Concentration of Xylazine in blood as determined by lab.

SECONDARY OUTCOMES:
Xylazine Strip Specificity and Sensitivity | 6 months
  Measuring Xylazine test strip specificity and sensitivity using excess urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Love, MD, MS, Principal Investigator — Icahn School of Medicine
Locations (2):
- United States (2):
  - NYC Health + Hospitals/Elmhurst, Elmhurst, New York
  - Icahn School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No
Not a clinical trial